CLINICAL TRIAL: NCT05577559
Title: Regional Analgesia Using Ultrasound-Guided Intermediate Cervical Plexus Block or Cervical Erector Spinae Block for Anterior Cervical Spine Surgery: A Randomized Trial
Brief Title: Ultrasound-Guided Intermediate Cervical Plexus or Cervical Erector Spinae Block for Anterior Cervical Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, Assistant professor of Anesthesia, Intensive Care and Pain Management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9790
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial cervical group (Active Comparator): patients will receive bilateral ultrasound guided intermediate cervical plexus block using 15 ml of bupivacaine 0.25% for each side.
  Interventions: Procedure: intermediate cervical plexus block
- Erector spinae group (Active Comparator): patients will receive bilateral ultrasound guided cervical erector spinae plane block using 15 ml of bupivacaine 0.25% for each side at the level of C6.
  Interventions: Procedure: Cervical Erector spinae block

INTERVENTIONS:
Procedure: intermediate cervical plexus block — patients will receive bilateral ultrasound guided intermediate cervical plexus block using 15 ml of bupivacaine 0.25% for each side.
  Arms: Superficial cervical group
Procedure: Cervical Erector spinae block — patients will receive bilateral ultrasound guided cervical erector spinae plane block using 15 ml of bupivacaine 0.25% for each side at the level of C6.
  Arms: Erector spinae group

SUMMARY:
• Neck pain and stiffness or sore throat, are common after anterior cervical spine surgery. Complications are rare but can be serious and even potentially life-threatening if they do occur. Rapid recovery and emergence from general anesthesia are important in cases of anterior cervical spine surgery.

DETAILED DESCRIPTION:
* Null hypothesis (H0): No difference between the regional analgesia effects of bilateral ultrasound-guided superficial cervical plexus block and bilateral cervical erector spinae block in patients undergoing anterior cervical spine surgery under general anesthesia.
* Alternative hypothesis (H1): There are differences between the regional analgesia effects of bilateral ultrasound-guided superficial cervical plexus block and bilateral cervical erector spinae block in

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age (21-60) years old.
* Both sex
* American Society of Anesthesiologist physical status I / II
* Elective anterior cervical spine surgery under general anesthesia.
* patient With Body Mass Index (BMI) (25-35kg/m²)

Exclusion Criteria:

* Local infection at site of puncture.
* Altered mental status.
* History of allergy to study drugs ( bupivacaine, fentanyl).
* Patients with chronic pain.
* Patients with severe hepatic or kidney impairment.
* Patients having a history of hematological disorders, including coagulation abnormality.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The time to first call to rescue analgesia | 24 hour postoperative
  The time to first call to rescue analgesia (nalbuphine) the time between the end of surgery to first report of postoperative pain. will be recorded.

SECONDARY OUTCOMES:
The total amount of nalbuphine | 24 hour postoperative
  The total amount of nalbuphine given to each patient during the first 24h of postoperative period will be recorded
Pain intensity | up to 24hs postoperative
  2. Pain intensity using Visual Analouge Scale (VAS) (11). A commonly used visual analog scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border. The patient is instructed to make a mark along the line to represent the intensity of pain currently being experienced. VAS score will be assessed at 30 minutes, 2hs, 4hs, 6hs, 12hs, and 24hs postoperative and IV increment of 15mg nalbuphine (rescue analgesic) will be given if VAS≥4.
Total intra-operative fentanyl consumption | intra-operative
  Total intra-operative fentanyl consumption by ug excluding induction dose.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, MD., Principal Investigator — Zagazig University, Faculty of Human Medicine
Locations (1):
- Faculty of Human Medicine, Zagazig University, Zagazig, Egypt

REFERENCES:
- [Derived] Kamel AAF, Fahmy AM, Fathi HM, Elmesallamy WAEA, Khalifa OYA. Regional analgesia using ultrasound-guided intermediate cervical plexus block versus cervical erector spinae block for anterior cervical spine surgery: a randomized trial. BMC Anesthesiol. 2024 Apr 22;24(1):153. doi: 10.1186/s12871-024-02533-6. PMID 38649826